CLINICAL TRIAL: NCT00478023
Title: A Randomized, Double-blind, Parallel-arm, Placebo- and Comparator- Controlled Trial of the Efficacy and Safety of Multiple Doses of Immediate-release (IR) CG5503 for Postoperative Pain Following Abdominal Hysterectomy
Brief Title: A Study to Evaluate the Efficacy and Safety of Tapentadol (CG5503) in the Treatment of Acute Pain After Abdominal Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 731200
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Hysterectomy; Postoperative
Keywords: Opioid; Central acting analgesic; Pain postoperative; Abdomen acute; CG5503 IR; Morphine; Placebo
MeSH Terms: conditions — Pain, Postoperative; Abdomen, Acute | interventions — Morphine; Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Morphine (Active Comparator)
  Interventions: Drug: Morphine
- Tapentadol 50 mg immediate release (Experimental)
  Interventions: Drug: CG5503 IR
- Tapentadol 75 mg immediate release (Experimental)
  Interventions: Drug: CG5503 IR
- Tapentadol 100 mg immediate release (Experimental)
  Interventions: Drug: CG5503 IR
- Matched placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine — 20 mg IR; 4 - 6 hourly; Total 72 hours
  Arms: Morphine
Drug: CG5503 IR — 50mg; 4 - 6 hourly; Total 72 hours
  Other Names: Tapentadol
  Arms: Tapentadol 50 mg immediate release
Drug: CG5503 IR — 75mg; 4 -6 hourly; Total 72 hours
  Other Names: Tapentadol
  Arms: Tapentadol 75 mg immediate release
Drug: CG5503 IR — 100mg, 4 - 6 hourly; Total 72 hours
  Other Names: Tapentadol
  Arms: Tapentadol 100 mg immediate release
Drug: Placebo — 4 - 6 hourly; Total 72 hours
  Arms: Matched placebo

SUMMARY:
The main objective of this study is to demonstrate the efficacy and safety of multiple-dose application of three different oral doses of CG5503 IR (tapentadol immediate release) compared to placebo in women undergoing abdominal hysterectomy.

DETAILED DESCRIPTION:
Subjects undergoing abdominal hysterectomy often experience moderate to severe acute pain post-surgery. Normally such pain is controlled when subjects receive repeated doses of opioid analgesics. However, opioid therapy is commonly associated with side effects such as nausea, vomiting, sedation, constipation, addiction, tolerance, and respiratory depression. Tapentadol (CG5503), a newly synthesized drug with an immediate release (IR) formulation, also acts as a centrally acting pain reliever but has a dual mode of action. The aim of this study is to investigate the effectiveness (level of pain control) and safety (side effects) of 3 dose levels of CG5503 IR compared with no drug (placebo) or one dose level of morphine (an opioid commonly used to treat post-surgical pain). This study is a randomized, double-blind (neither investigator nor patient will know which treatment was received), active- and placebo-controlled, parallel-group, multicenter study to evaluate the treatment of acute pain after abdominal hysterectomy. The study will include a blinded 72 hour in-patient phase immediately following hysterectomy, during which subjects will be treated with either 50-, 75-, or 100-mg CG5503 IR, a matched placebo, or 20-mg morphine, and pain relief will be periodically assessed. Assessments of pain relief include the pain intensity numeric rating scale (PI), pain relief numeric rating scale (PAR), and patient global impression of change scale (PGIC). Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. Venous blood samples will be collected for the determination of serum concentrations of CG5503 and morphine. The alternative study hypothesis is that at least 1 dose strength of CG5503 will be different from placebo in controlling pain at 24 hours (using the mean SPID at 24 hours).

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 80 years of age;
* Scheduled to undergo an abdominal hysterectomy with or without bilateral salpingo-oophorectomy due to uterine leiomyomas, or dysfunctional uterine bleeding or endometrial hyperplasia;
* Anesthesiological and surgical procedures performed according to protocol;
* Moderate or severe baseline pain following hysterectomy on a Verbal Rating Scale (VRS) within 6 hours following the last possible application of morphine subcutaneous;
* Pain following hysterectomy of at least 4 on an 11-point Numeric Rating Scale (NRS) within 6 hours following the last possible application of morphine subcutaneous;
* American Society of Anesthesiologists (ASA) classification I-III.

Exclusion Criteria:

* Vaginal hysterectomy;
* Ongoing or known history of painful endometriosis;
* Known or suspected chronic pelvic pain syndrome;
* Previous abdominal or pelvic open surgery;
* History of seizure disorder or epilepsy;
* History of alcohol or drug abuse;
* Evidence of active infections that may spread to other areas of the body;
* severely impaired renal function, moderately or severely impaired hepatic function,
* Allergy or hypersensitivity to oxycodone, morphine, fentanyl hydromorphone, heparin, or any compound planned to be used during the anesthesia;
* Serious complication during surgery and up to randomization;
* Pre-operative use within 12hours prior to surgery or peri-operative use of non-steroidal anti-inflammatory drugs (NSAIDs);
* Treated regularly with opioid analgesic or non-steroidal anti-inflammatory drugs (NSAIDs) within 30 days prior to screening;

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Rechberger, Prof., Principal Investigator — Samodzielny Publiczny Szpital
Locations (52):
- Hungary (4):
  - Site 13, Békéscsaba
  - Site 14, Debrecen
  - Site 15, Komárom
  - Site 12, Nyíregyháza
- Latvia (4):
  - Site 16, Riga
  - Site 17, Riga
  - Site 18, Riga
  - Site 19, Riga
- Poland (10):
  - Site 27, Katowice
  - Site 23, Krakow
  - Site 24, Lodz
  - Site 66, Lodz
  - Site 22, Lublin
  - Site 25, Lublin
  - Site 26, Ruda Śląska
  - Site 20, Warsaw
  - Site 21, Warsaw
  - Site 28, Wroclaw
- Romania (12):
  - Site 33, Brasov
  - Site 78, Brasov
  - Site 29, Bucharest
  - Site 30, Bucharest
  - Site 31, Bucharest
  - Site 32, Bucharest
  - Site 34, Bucharest
  - Site 35, Bucharest
  - Site 36, Bucharest
  - Site 76, Bucharest
  - Site 75, Craiova
  - Site 61, Ploieşti
- Russia (7):
  - Site 71, Belgorod
  - Site 37, Moscow
  - Site 38, Moscow
  - Site 44, Moscow
  - Site 73, Moscow
  - Site 42, Saint Petersburg
  - Site 43, Saint Petersburg
- Serbia (4):
  - Site 45, Belgrade
  - Site 47, Belgrade
  - Site 46, Kragujevac
  - Site 70, Novi Sad
- Slovakia (5):
  - Site 48, Banská Bystrica
  - Site 51, Bratislava
  - Site 52, Bratislava
  - Site 62, Košice
  - Site 50, Martin
- Site 53, Maribor, Slovenia
- Ukraine (5):
  - Site 64, Donetsk
  - Site 55, Kiev
  - Site 56, Kiev
  - Site 58, Kiev
  - Site 67, Zaporizhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this in-patient, multicenter study occurred between 19 May 2007 and 11 Mar 2008.
Pre-assignment Details: This trial consisted of 5 periods: a Screening (Day -28 to Day -4 to the Pre-operative Visit) a Surgical (Day -1 to 1), a Postoperative Qualification, a Double-blind Treatment(Day 1-4) and a Follow-up Period (4-14 days after the double-blind treatment). The results refer to randomized subjects.
Groups:
- Morphine: Morphine IR 20mg 4-6 hourly
- CG5503 50mg: CG5503 IR 50mg 4 to 6 hourly
- CG5503 75mg: CG5503 IR 75mg 4 to 6 hourly
- CG5503 100mg: CG5503 IR 100mg 4 to 6 hourly
- Placebo: Matched Placebo 4 to 6 hourly
Period: Overall Study
Arm/Group | Morphine | CG5503 50mg | CG5503 75mg | CG5503 100mg | Placebo
Started | 170 | 168 | 171 | 176 | 169
Completed | 135 | 144 | 151 | 146 | 114
Not Completed | 35 | 24 | 20 | 30 | 55
Not completed — Adverse Event | 11 | 7 | 8 | 14 | 6
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 11 | 10 | 4 | 5 | 41
Not completed — Lost to Follow-up | 3 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 4 | 5
Not completed — Lack of pain, Technical difficulties | 7 | 3 | 5 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | CG5503 50mg | CG5503 75mg | CG5503 100mg | Placebo | Total
Number analyzed (Participants) | 170 | 168 | 171 | 176 | 169 | 854
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 165 | 166 | 170 | 173 | 166 | 840
  >=65 years | 5 | 2 | 1 | 3 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (6.75) | 47.0 (5.56) | 47.1 (5.37) | 47.5 (6.43) | 47.2 (5.83) | 47.5 (6.03)
Sex/Gender, Customized [Number; unit: participants]
  Female | 170 | 168 | 171 | 176 | 169 | 854
Region of Enrollment [Number; unit: participants]
  Serbia | 15 | 15 | 16 | 16 | 15 | 77
  Hungary | 5 | 6 | 5 | 5 | 4 | 25
  Slovakia | 25 | 25 | 25 | 25 | 24 | 124
  Poland | 36 | 36 | 34 | 37 | 36 | 179
  Ukraine | 14 | 11 | 14 | 14 | 13 | 66
  Romania | 34 | 33 | 34 | 36 | 35 | 172
  Russian Federation | 21 | 21 | 21 | 22 | 22 | 107
  Latvia | 20 | 21 | 22 | 21 | 20 | 104

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Differences Relative to the Baseline Pain Intensity.
Description: Pain Intensity assessed at predefined time points over a 24 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Differences calculated as [baseline-post baseline] at each predefined time point. The theoretical maximum range of Sum of pain intensity differences (SPID24) is from -240 (indicative of an increase in pain) to 240 (indicative of a decrease in pain, assuming patients start with a baseline value of 10 and all subsequent values will be 0).
Time Frame: Baseline to 24 hours after first intake of study drug
Population: Intention to Treat (ITT) and Last Observation Carried Forward (LOCF), i.e. all randomized subjects who received any amount of Investigational Medicinal Product (IMP = study drug) and had a non missing baseline pain assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Morphine | CG5503 50mg | CG5503 75mg | CG5503 100mg | Placebo
Number analyzed (Participants) | 164 | 163 | 167 | 172 | 166
units on scale | 48.8 (41.0) | 49.0 (39.87) | 52.4 (41.85) | 52.9 (40.95) | 29.0 (44.98)
Statistical Analysis 1: Comparison: CG5503 50mg vs Placebo; The null hypothesis is that all CG5503 IR dose groups are equal to the placebo group based on the mean sum of pain intensity difference at 24 hours (SPID24). The alternative hypothesis is that at least one CG5503 IR dose group is different from the placebo group based on the mean SPID24; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted. The Hochberg procedure used for multiplicity comparisons; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean difference = 18.1, 95% CI [10.9 to 25.3] — Only pain intensity assessments collected prior to the first dose of any additional analgesic medication considered. Afterwards LOCF used
Statistical Analysis 2: Comparison: CG5503 75mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted. The Hochberg procedure used for multiplicity comparisons; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean difference = 20.8, 95% CI [13.7 to 28.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: CG5503 100mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted. The Hochberg procedure used for multiplicity comparisons; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean difference = 23.3, 95% CI [16.3 to 30.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Morphine vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustment used; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean difference = 20.6, 95% CI [13.4 to 27.8] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Sum of Pain Intensity Differences Relative to the Baseline Pain Intensity
Description: Pain Intensity assessed at predefined time points over a 48 hour period using an 11-point Numeric Rating Scale (NRS) where a score of zero indicates "no pain" and a score of ten indicates "pain as bad as you can imagine". Differences calculated as [baseline-post baseline] at each predefined time point. The theoretical maximum range of Sum of pain intensity differences (SPID48) is from -480 (indicative of an increase in pain) to 480 (indicative of a decrease in pain, assuming patients start with a baseline value of 10 and all subsequent values will be 0).
Time Frame: Baseline value to 48 hours after first study drug intake.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Morphine | CG5503 50mg | CG5503 75mg | CG5503 100mg | Placebo
Number analyzed (Participants) | 164 | 163 | 167 | 172 | 166
units on scale | 116.6 (87.10) | 112.4 (87.32) | 120.6 (87.35) | 123.5 (83.50) | 71.1 (101.17)
Statistical Analysis 1: Comparison: CG5503 50mg vs Placebo; The null hypothesis is that all CG5503 IR dose groups are equal to the placebo group based on the mean sum of pain intensity difference at 48 hours (SPID48). The alternative hypothesis is that at least one CG5503 IR dose group is different from the placebo group based on the mean SPID48; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted. The Hochberg procedure used for multiplicity comparisons; ANCOVA with treatment and centre as fixed effects and baseline pain as covariate; Least square mean difference = 37.1, 95% CI [21.6 to 52.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CG5503 75mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted. The Hochberg procedure used for multiplicity comparisons; ANCOVA with treatment and centre as fixed effects and baseline pain as covariates; Least square mean difference = 44.0, 95% CI [28.6 to 59.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: CG5503 100mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Adjusted. The Hochberg procedure used for multiplicity comparisons; Least square mean difference = 51.4, 95% CI [36.1 to 66.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Morphine vs Placebo; Null hypothesis of no treatment difference; Test type: Superiority or Other; p < 0.0001, ANCOVA — No multiplicity adjustment; ANCOVA with treatment and centre as fixed effects and baseline pain as a covariate; Least square mean difference = 46.9, 95% CI [31.4 to 62.4] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events are reported.
Arm/Group | Morphine | CG5503 50mg | CG5503 75mg | CG5503 100mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/170 | 0/168 | 0/171 | 1/176 | 0/169
Other Adverse Events (participants affected / at risk) | 99/170 | 84/168 | 96/171 | 106/176 | 88/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=170) | CG5503 50mg (N=168) | CG5503 75mg (N=171) | CG5503 100mg (N=176) | Placebo (N=169)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (N=170) | CG5503 50mg (N=168) | CG5503 75mg (N=171) | CG5503 100mg (N=176) | Placebo (N=169)
Nausea (Gastrointestinal disorders) | 31 | 23 | 33 | 31 | 21
Constipation (Gastrointestinal disorders) | 13 | 11 | 10 | 15 | 9
Vomiting (Gastrointestinal disorders) | 11 | 12 | 13 | 20 | 4
Flatulence (Gastrointestinal disorders) | 14 | 12 | 12 | 14 | 11
Dizziness (Nervous system disorders) | 7 | 9 | 7 | 21 | 8
Somnolence (Nervous system disorders) | 14 | 6 | 9 | 13 | 4
Headache (Nervous system disorders) | 9 | 5 | 10 | 10 | 11
Pyrexia (General disorders) | 15 | 15 | 16 | 13 | 16
Body temperature increased (Investigations) | 4 | 6 | 7 | 1 | 10
Postoperative anemia (Injury, poisoning and procedural complications) | 8 | 5 | 5 | 4 | 10

LIMITATIONS AND CAVEATS:
Approval to conduct the trial was obtained in Slovenia. No Slovenian subjects were exposed to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Grünenthal GmbH reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither Grünenthal nor the coordinating Investigator/Investigator has the right to prohibit publication unless publication can be shown to affect possible patent rights.